CLINICAL TRIAL: NCT00084981
Title: A Phase I Study of Decitabine in Combination With Valproic Acid in Patients With Non-Small Cell Lung Cancer
Brief Title: Decitabine and Valproic Acid in Treating Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01451; NCI-2012-01451 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-6237; OSU-2003C0087; OSU-0346; CDR0000367115; OSU 0346 (Other: Ohio State University Medical Center); 6237 (Other: CTEP); U01CA076576 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Decitabine; Valproic Acid

ARMS (1):
- Treatment (decitabine, valproic acid) (Experimental): Patients receive decitabine IV over 1 hour on days 1-10 and oral valproic acid three times daily on days 5-21. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of decitabine and valproic acid until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. After the MTD is determined, an additional 6 patients are treated at that dose.
  Interventions: Drug: decitabine; Drug: valproic acid; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Drug: valproic acid — Given PO
  Other Names: Alti-Valproic; Depakene; Novo-Valproic; VA
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of decitabine and valproic acid in treating patients with non-small cell lung cancer. Drugs used in chemotherapy, such as decitabine and valproic acid, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of decitabine and valproic acid in patients with non-small cell lung cancer.

II. Determine the recommended phase II dose of this regimen in these patients.

SECONDARY OBJECTIVES:

I. Determine the ability of this regimen to lead to biological changes in tumor and surrogate tissues in these patients, including hypomethylation of target genes known to be methylated in NSCLC (CDKN2, APC, BMP3B, CDH1 and RASSF1A) in biopsy specimens and surrogate tissues (peripheral blood mononuclear cells [PBMC] and plasma/serum DNA); acetylation and methylation changes in histones from tumor and surrogate tissues (PBMC and oral epithelial cells); inhibition of histone deacetylase (HDAC) activity in peripheral blood; pharmacokinetic analysis of Decitabine and Valproic Acid; DNA methyltransferase 1 (DNMT1) protein loss in PBMC and buccal cells; response of hemoglobin F in patients with non-hematologic conditions to DNMT and HDAC inhibition; and preliminary evidence of antitumor activity in non-small cell lung cancer.

OUTLINE: This is a dose-escalation study.

Patients receive decitabine IV over 1 hour on days 1-10 and oral valproic acid three times daily on days 5-21. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of decitabine and valproic acid until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. After the MTD is determined, an additional 6 patients are treated at that dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer
* Tumor accessible to biopsy by bronchoscopy, through surface biopsy (e.g., skin punch biopsy for skin/subcutaneous metastasis) or through CT scan guidance
* Not eligible for curative surgery, chemotherapy, radiotherapy, or multimodality treatment options
* No uncontrolled brain metastases

  * Controlled brain metastases allowed provided patient has no neurologic deterioration when off steroids; has completed prior radiotherapy or other treatments; has fully recovered from prior treatment; and does not require anticonvulsants
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 12 weeks
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* WBC > 3,000/mm^3
* AST and ALT =< 2.5 times upper limit of normal (ULN)
* Bilirubin =< 1.5 times ULN
* Creatinine =< 1.5 times ULN
* Creatinine clearance >= 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction to compounds of similar chemical or biological composition to decitabine, valproic acid, or other study agents
* No other concurrent uncontrolled illness
* No ongoing or active infection requiring antibiotics
* No history of seizures requiring anticonvulsants
* No medical problem that would preclude study participation
* No psychiatric illness or social situation that would preclude study compliance
* No other active malignancy except non-melanoma skin cancer or carcinoma in situ of the cervix
* No concurrent prophylactic growth factors (e.g., filgrastim [G-CSF] or epoetin alfa)
* No more than 3 prior chemotherapy regimens
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior definitive radiotherapy to the chest allowed

  * Clinical (radiographic or other) evidence of tumor progression for previously irradiated indicator lesion in the chest
* More than 2 weeks since prior radiotherapy and recovered
* No concurrent palliative radiotherapy
* Prior curative or palliative intent surgery allowed
* At least 2 weeks since prior surgery and recovered
* At least 4 weeks since prior photodynamic therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer agents or therapies
* No other concurrent investigational agents
* No concurrent administration of any of the following medications:

  * Aspirin

    * Chronic low-dose (=< 81 mg/day) aspirin allowed
  * Felbamate
  * Rifampin
  * Amitriptyline
  * Nortriptyline
  * Carbamazepine
  * Clonazepam
  * Diazepam
  * Ethosuximide
  * Lamotrigine
  * Phenobarbital
  * Barbiturates
  * Primidone
  * Phenytoin
  * Zidovudine
* No concurrent divalproex sodium
* Concurrent gabapentin for neuropathic pain allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-04; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
MTD, defined as dose in which fewer than 1/3 or 2/6 patients experience DLT | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Otterson, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States